CLINICAL TRIAL: NCT04967443
Title: A 2 COHORT, SINGLE DOSE, OPEN-LABEL, RANDOMIZED, PIVOTAL BIOEQUIVALENCE STUDY TO QUALIFY MANUFACTURING SITE TRANSFER FROM BARCELONETA TO ASCOLI FOR PRAZOSIN HYDROCHLORIDE CAPSULES IN HEALTHY ADULT PARTICIPANTS UNDER FASTED CONDITIONS
Brief Title: Pivotal Bioequivalence Study to Qualify Manufacturing Site Transfer for Prazosin Hydrochloride Capsules
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: A0281006
Record Dates: First submitted 2021-07-08; First posted 2021-07-19 (Actual); Results first posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-01

CONDITIONS: Hypertension; Heart Failure
MeSH Terms: conditions — Hypertension; Heart Failure | interventions — Prazosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Prazosin Hydrochloride (HCL) 2 milligram (mg) capsule Barceloneta site (Active Comparator): One 2 mg capsule manufactured at the current site, Barceloneta
  Interventions: Drug: Prazosin HCl 2mg
- Prazosin HCL 2 mg capsule Ascoli site (Experimental): One 2 mg capsule manufactured at the proposed site (Ascoli)
  Interventions: Drug: Prazosin HCl 2mg
- Prazosin HCL 1 mg capsule Ascoli site (Experimental): Two 1 mg capsule manufactured at the proposed site, Ascoli
  Interventions: Drug: Prazosin HCl 1 mg
- Prazosin HCL 5 mg capsule Barceloneta site (Active Comparator): One 5 mg capsule manufactured at the current site, Barceloneta
  Interventions: Drug: Prazosin HCl 5 mg
- Prazosin HCL 1 x 5 mg capsule Ascoli site (Active Comparator): One 5 mg capsule manufactured at the proposed site, Ascoli
  Interventions: Drug: Prazosin HCl 5 mg

INTERVENTIONS:
Drug: Prazosin HCl 2mg — Prazosin HCL 1 X 2 mg capsule.
  Other Names: Minipress 2 mg capsule.
  Arms: Prazosin HCL 2 mg capsule Ascoli site; Prazosin Hydrochloride (HCL) 2 milligram (mg) capsule Barceloneta site
Drug: Prazosin HCl 1 mg — Prazosin HCl 2 X 1 mg capsule.
  Other Names: Minipress 1 mg capsule.
  Arms: Prazosin HCL 1 mg capsule Ascoli site
Drug: Prazosin HCl 5 mg — Prazosin HCL 1 X 5 mg capsule.
  Other Names: Minipress 5 mg capsule.
  Arms: Prazosin HCL 1 x 5 mg capsule Ascoli site; Prazosin HCL 5 mg capsule Barceloneta site

SUMMARY:
Prazosin hydrochloride (HCl) is an oral anti-hypertensive indicated for the treatment of primary and secondary hypertension and heart failure. Pfizer Inc. is the marketing authorization holder for prazosin HCl oral capsules and intended to transfer drug product manufacturing operations from Pfizer, Barceloneta Puerto Rico to Pfizer Pharmaceutical, Ascoli, Italy. To support the manufacturer site transfer and process changes, this bioequivalence (BE) study is being conducted.

This study will be a 2 Cohort, open-label, randomized, single dose study in healthy adult male and/or female participants. Cohort 1 will be crossover with 3 treatments, 3 periods, 6 sequences. Cohort 2 will be crossover with 2 treatments, 2 periods, 2 sequences. Primary objective of this study is demonstrate bioequivalence between prazosin HCl 1, 2 and 5 mg capsules manufactured at Ascoli versus prazosin HCl 2 and 5 mg capsules manufactured at Barceloneta under fasting conditions in healthy adult participants. Approximately 36 participants will be enrolled in each Cohort 1 and Cohort 2.

Pharmacokinetic and statistical analysis will be performed for prazosin. Data from 2 Cohorts will be analyzed separately. The PK parameters area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration (AUClast), and from time zero extrapolated to infinite time (AUCinf), maximum plasma concentration (Cmax), time to first occurrence of Cmax (Tmax), and terminal phase elimination half-life (t½) will be summarized descriptively by analyte and treatment.

For primary objective, bioequivalence of the Test treatment relative to Reference treatment will be concluded if the 90% confidence intervals (CI) for the ratio of adjusted geometric means of Test treatments relative to Reference treatment for AUCinf (if data permit), AUClast and Cmax, fall wholly within (80%, 125%).

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18 to 55 years of age, inclusive, at the time of signing the Informed Consent Document (ICD).
* Male and female participants who are overtly healthy as determined by medical evaluation including medical history, full physical examination, vital signs, 12-lead electrocardiogram (ECG), and/or clinical laboratory tests.
* Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations , and other study procedures.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb).
* Capable of giving signed informed consent as described in Appendix 1, which includes compliance with the requirements and restrictions listed in the ICD and in this protocol.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease.
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* History of Human Immunodeficiency Virus (HIV) infection, hepatitis B, or hepatitis C; positive testing for HIV, hepatitis B surface antigen (HBsAg), hepatitis B surface antibody (HBsAb) or hepatitis C antibody (HCVAb). Hepatitis B vaccination is allowed.
* Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half lives (whichever is longer) prior to the first dose of study intervention.
* A positive urine drug test.
* Screening supine blood pressure (BP) ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), following at least 5 minutes of supine rest.
* Baseline standard 12 lead ECG that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results.
* Participants with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study specific laboratory and confirmed by a single repeat test, if deemed necessary:
* aspartate aminotransferase (AST) or alanine aminotransferase (ALT) level ≥1.5 × upper limit of normal (ULN);
* Total bilirubin level ≥1.5 × ULN; participants with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is ≤ ULN.
* History of alcohol abuse or binge drinking and/or any other illicit drug use or dependence within 6 months of Screening.
* Use of tobacco or nicotine containing products in excess of the equivalent of 5 cigarettes per day. For chewing tobacco, one chew is equivalent to approximately 2 to 3 cigarettes, so participants would be limited to 2 or less chews per day.
* History of sensitivity to prazosin hydrochloride or any of the components in the formulation of the study products.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2021-09-22 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Clinical Trials of Texas, LLC, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A0281006

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 72 participants were enrolled in the study and both cohorts (2 cohorts in total) enrolled 36 particpants.
Groups:
- Prazosin HCL 1x2 mg (Barceloneta) => Prazosin HCL 1x2 mg (Ascoli) => Prazosin HCL 2x1 mg (Ascoli); Prazosin HCL 1x2 mg (Barceloneta) => Prazosin HCL 2x1 mg (Ascoli) => Prazosin HCL 1x2 mg (Ascoli); Prazosin HCL 1x2 mg (Ascoli) => Prazosin HCL 1x2 mg (Barceloneta) => Prazosin HCL 2x1 mg (Ascoli); Prazosin HCL 1x2 mg (Ascoli) => Prazosin HCL 2x1 mg (Ascoli) => Prazosin HCL 1x2 mg (Barceloneta); Prazosin HCL 2x1 mg (Ascoli) => Prazosin HCL 1x2 mg (Barceloneta) => Prazosin HCL 1x2 mg (Ascoli); Prazosin HCL 2x1 mg (Ascoli) => Prazosin HCL 1x2 mg (Ascoli) => Prazosin HCL 1x2 mg (Barceloneta): Cohort 1, Prazosin HCL were given to participants under fasted conditions. There's an at least 7-day washout period between treatment periods.
- Prazosin HCL 1x5 mg (Barceloneta) => Prazosin HCL 1x5 mg (Ascoli); Prazosin HCL 1x5 mg (Ascoli) => Prazosin HCL 1x5 mg (Barceloneta): Cohort 2, Prazosin HCl were given to participants under fasted conditions. There's an at least 7-day washout period between treatment periods.
Period: Screening
Arm/Group | Prazosin HCL 1x2 mg (Barceloneta) => Prazosin HCL 1x2 mg (Ascoli) => Prazosin HCL 2x1 mg (Ascoli) | Prazosin HCL 1x2 mg (Barceloneta) => Prazosin HCL 2x1 mg (Ascoli) => Prazosin HCL 1x2 mg (Ascoli) | Prazosin HCL 1x2 mg (Ascoli) => Prazosin HCL 1x2 mg (Barceloneta) => Prazosin HCL 2x1 mg (Ascoli) | Prazosin HCL 1x2 mg (Ascoli) => Prazosin HCL 2x1 mg (Ascoli) => Prazosin HCL 1x2 mg (Barceloneta) | Prazosin HCL 2x1 mg (Ascoli) => Prazosin HCL 1x2 mg (Barceloneta) => Prazosin HCL 1x2 mg (Ascoli) | Prazosin HCL 2x1 mg (Ascoli) => Prazosin HCL 1x2 mg (Ascoli) => Prazosin HCL 1x2 mg (Barceloneta) | Prazosin HCL 1x5 mg (Barceloneta) => Prazosin HCL 1x5 mg (Ascoli) | Prazosin HCL 1x5 mg (Ascoli) => Prazosin HCL 1x5 mg (Barceloneta)
Started | 6 | 6 | 6 | 6 | 6 | 6 | 18 | 18
Completed | 6 | 6 | 6 | 6 | 6 | 6 | 18 | 18
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Open Label Treatment
Arm/Group | Prazosin HCL 1x2 mg (Barceloneta) => Prazosin HCL 1x2 mg (Ascoli) => Prazosin HCL 2x1 mg (Ascoli) | Prazosin HCL 1x2 mg (Barceloneta) => Prazosin HCL 2x1 mg (Ascoli) => Prazosin HCL 1x2 mg (Ascoli) | Prazosin HCL 1x2 mg (Ascoli) => Prazosin HCL 1x2 mg (Barceloneta) => Prazosin HCL 2x1 mg (Ascoli) | Prazosin HCL 1x2 mg (Ascoli) => Prazosin HCL 2x1 mg (Ascoli) => Prazosin HCL 1x2 mg (Barceloneta) | Prazosin HCL 2x1 mg (Ascoli) => Prazosin HCL 1x2 mg (Barceloneta) => Prazosin HCL 1x2 mg (Ascoli) | Prazosin HCL 2x1 mg (Ascoli) => Prazosin HCL 1x2 mg (Ascoli) => Prazosin HCL 1x2 mg (Barceloneta) | Prazosin HCL 1x5 mg (Barceloneta) => Prazosin HCL 1x5 mg (Ascoli) | Prazosin HCL 1x5 mg (Ascoli) => Prazosin HCL 1x5 mg (Barceloneta)
Started | 6 | 6 | 6 | 6 | 6 | 6 | 18 | 18
Completed | 5 | 5 | 5 | 5 | 6 | 5 | 16 | 15
Not Completed | 1 | 1 | 1 | 1 | 0 | 1 | 2 | 3
Not completed — Death | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 3
Period: Follow-Up
Arm/Group | Prazosin HCL 1x2 mg (Barceloneta) => Prazosin HCL 1x2 mg (Ascoli) => Prazosin HCL 2x1 mg (Ascoli) | Prazosin HCL 1x2 mg (Barceloneta) => Prazosin HCL 2x1 mg (Ascoli) => Prazosin HCL 1x2 mg (Ascoli) | Prazosin HCL 1x2 mg (Ascoli) => Prazosin HCL 1x2 mg (Barceloneta) => Prazosin HCL 2x1 mg (Ascoli) | Prazosin HCL 1x2 mg (Ascoli) => Prazosin HCL 2x1 mg (Ascoli) => Prazosin HCL 1x2 mg (Barceloneta) | Prazosin HCL 2x1 mg (Ascoli) => Prazosin HCL 1x2 mg (Barceloneta) => Prazosin HCL 1x2 mg (Ascoli) | Prazosin HCL 2x1 mg (Ascoli) => Prazosin HCL 1x2 mg (Ascoli) => Prazosin HCL 1x2 mg (Barceloneta) | Prazosin HCL 1x5 mg (Barceloneta) => Prazosin HCL 1x5 mg (Ascoli) | Prazosin HCL 1x5 mg (Ascoli) => Prazosin HCL 1x5 mg (Barceloneta)
Started (Participants who entered the follow-up period is calculated as participants who had open-label treatments as follow-up occurred 28-35 days from last dose of study treatment administration.) | 6 | 6 | 6 | 6 | 6 | 6 | 18 | 18
Completed | 5 | 5 | 5 | 4 | 6 | 5 | 16 | 15
Not Completed | 1 | 1 | 1 | 2 | 0 | 1 | 2 | 3
Not completed — Death | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1: Male: Male participants enrolled to the cohort 1 of the study.
- Cohort 1: Female: Female participants enrolled to the cohort 1 of the study.
- Cohort 2: Male: Male participants enrolled to the cohort 2 of the study.
- Cohort 2: Female: Female participants enrolled to the cohort 2 of the study.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Male | Cohort 1: Female | Cohort 2: Male | Cohort 2: Female | Total
Number analyzed (Participants) | 24 | 12 | 20 | 16 | 72
Age, Customized [Number; unit: Participants]
  <18 years | 0 | 0 | 0 | 0 | 0
  18-44 years | 16 | 7 | 18 | 10 | 51
  45-64 years | 8 | 5 | 2 | 6 | 21
  ≥65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 12 | 0 | 16 | 28
  Male | 24 | 0 | 20 | 0 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 4 | 8 | 9 | 32
  Not Hispanic or Latino | 13 | 8 | 12 | 7 | 40
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 2 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1
  Black or African American | 8 | 1 | 5 | 4 | 18
  White | 16 | 8 | 13 | 12 | 49
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Last Quantifiable Concentration (AUClast) of Prazosin
Time Frame: 0 (pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 10, 12, 24 hours post-dose on Day 1 of each period
Population: The AUClast analysis population is defined as all participants randomized and treated who had at least 1 of the PK parameters of primary interest in at least 1 treatment period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Groups:
- Prazosin HCL 1x2 mg (Barceloneta): Cohort 1, Prazosin HCl 2 mg capsules, manufactured at Pfizer Pharmaceutical, Barceloneta, Puerto Rico, were given to participants under fasted conditions.
- Prazosin HCL 1x2 mg (Ascoli): Cohort 1, Prazosin HCl 2 mg capsules, manufactured at Pfizer Pharmaceutical, Ascoli, Italy, were given to participants under fasted conditions.
- Prazosin HCL 2x1 mg (Ascoli): Cohort 1, Prazosin HCl 1 mg capsules, manufactured at Pfizer Pharmaceutical, Ascoli, Italy, were given to participants under fasted conditions.
- Prazosin HCL 1x5 mg (Barceloneta): Cohort 2, Prazosin HCl 5 mg capsules, manufactured at Pfizer Pharmaceutical, Barceloneta, Puerto Rico, were given to participants under fasted conditions.
- Prazosin HCL 1x5 mg (Ascoli): Cohort 2, Prazosin HCl 5 mg capsules, manufactured at Pfizer Pharmaceutical, Ascoli, Italy, were given to participants under fasted conditions.
Arm/Group | Prazosin HCL 1x2 mg (Barceloneta) | Prazosin HCL 1x2 mg (Ascoli) | Prazosin HCL 2x1 mg (Ascoli) | Prazosin HCL 1x5 mg (Barceloneta) | Prazosin HCL 1x5 mg (Ascoli)
Number analyzed (Participants) | 34 | 33 | 32 | 33 | 34
nanogram*hour per milliliter (ng*hr/mL) | 85.77 (34) | 88.37 (31) | 92.39 (34) | 192.3 (147) | 252.2 (37)
Statistical Analysis 1: Comparison: Prazosin HCL 1x2 mg (Ascoli); Test: Prazosin HCL 1x2 mg (Ascoli); Reference: Prazosin HCL 1x2 mg (Barceloneta); Test type: Equivalence — Bioequivalence will be demonstrated if the estimated 90% confidence interval for the ratios (Test/Reference) of adjusted geometric means for AUClast and Cmax fall entirely within (80%, 125%); Mixed Models Analysis; Ratio of adjusted geometric means = 102.10, 90% CI 2-sided [96.14 to 108.43]
Statistical Analysis 2: Comparison: Prazosin HCL 2x1 mg (Ascoli); Test: Prazosin HCL 2x1 mg (Ascoli); Reference: Prazosin HCL 1x2 mg (Barceloneta); Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; Ratio of adjusted geometric means = 104.87, 90% CI 2-sided [98.68 to 111.44]
Statistical Analysis 3: Comparison: Prazosin HCL 1x5 mg (Barceloneta) vs Prazosin HCL 1x5 mg (Ascoli); Test: Prazosin HCL 1x5 mg (Ascoli); Reference: Prazosin HCL 1x5 mg (Barceloneta); Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; Ratio of adjusted geometric means = 104.45, 90% CI 2-sided [99.58 to 109.55]

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Prazosin
Time Frame: 0 (pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 10, 12, 24 hours post-dose on Day 1 of each period
Population: The Cmax analysis population is defined as all participants randomized and treated who had at least 1 of the PK parameters of primary interest in at least 1 treatment period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Prazosin HCL 1x2 mg (Barceloneta) | Prazosin HCL 1x2 mg (Ascoli) | Prazosin HCL 2x1 mg (Ascoli) | Prazosin HCL 1x5 mg (Barceloneta) | Prazosin HCL 1x5 mg (Ascoli)
Number analyzed (Participants) | 34 | 33 | 33 | 33 | 34
nanogram per milliliter (ng/mL) | 14.82 (49) | 17.04 (36) | 19.20 (37) | 30.91 (143) | 38.69 (132)
Statistical Analysis 1: Comparison: Prazosin HCL 1x2 mg (Ascoli); Test: Prazosin HCL 1x2 mg (Ascoli); Reference: Prazosin HCL 1x2 mg (Barceloneta); Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; Ratio of adjusted geometric means = 113.96, 90% CI 2-sided [102.79 to 126.34]
Statistical Analysis 2: Comparison: Prazosin HCL 2x1 mg (Ascoli); Test: Prazosin HCL 2x1 mg (Ascoli); Reference: Prazosin HCL 1x2 mg (Barceloneta); Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; Ratio of adjusted geometric means = 126.83, 90% CI 2-sided [114.32 to 140.70]
Statistical Analysis 3: Comparison: Prazosin HCL 1x5 mg (Barceloneta) vs Prazosin HCL 1x5 mg (Ascoli); Test: Prazosin HCL 1x5 mg (Ascoli); Reference: Prazosin HCL 1x5 mg (Barceloneta); Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; Ratio of adjusted geometric means = 118.07, 90% CI 2-sided [106.46 to 130.94]

3. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Extrapolated Infinite Time (AUCinf) of Prazosin
Time Frame: 0 (pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 10, 12, 24 hours post-dose on Day 1 of each period
Population: The AUCinf analysis population is defined as all participants randomized and treated who had at least 1 of the PK parameters of secondary interest in at least 1 treatment period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Prazosin HCL 1x2 mg (Barceloneta) | Prazosin HCL 1x2 mg (Ascoli) | Prazosin HCL 2x1 mg (Ascoli) | Prazosin HCL 1x5 mg (Barceloneta) | Prazosin HCL 1x5 mg (Ascoli)
Number analyzed (Participants) | 31 | 32 | 31 | 32 | 33
ng*hr/mL | 89.10 (33) | 90.28 (31) | 93.01 (31) | 236.7 (37) | 259.0 (37)
Statistical Analysis 1: Comparison: Prazosin HCL 1x2 mg (Ascoli); Test: Prazosin HCL 1x2 mg (Ascoli); Reference: Prazosin HCL 1x2 mg (Barceloneta); Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; Ratio of adjusted geometric means = 100.91, 90% CI 2-sided [94.92 to 107.27]
Statistical Analysis 2: Comparison: Prazosin HCL 2x1 mg (Ascoli); Test: Prazosin HCL 2x1 mg (Ascoli); Reference: Prazosin HCL 1x2 mg (Barceloneta); Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; Ratio of adjusted geometric means = 102.08, 90% CI 2-sided [95.97 to 108.57]
Statistical Analysis 3: Comparison: Prazosin HCL 1x5 mg (Barceloneta) vs Prazosin HCL 1x5 mg (Ascoli); Test: Prazosin HCL 1x5 mg (Ascoli); Reference: Prazosin HCL 1x5 mg (Barceloneta); Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; Ratio of adjusted geometric means = 104.04, 90% CI 2-sided [99.09 to 109.23]

4. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Prazosin
Time Frame: 0 (pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 10, 12, 24 hours post-dose on Day 1 of each period
Population: The Tmax analysis population is defined as all participants randomized and treated who had at least 1 of the PK parameters of secondary interest in at least 1 treatment period.
Measure: Median (Full Range); unit: hr
Arm/Group | Prazosin HCL 1x2 mg (Barceloneta) | Prazosin HCL 1x2 mg (Ascoli) | Prazosin HCL 2x1 mg (Ascoli) | Prazosin HCL 1x5 mg (Barceloneta) | Prazosin HCL 1x5 mg (Ascoli)
Number analyzed (Participants) | 33 | 33 | 33 | 33 | 34
hr | 2.00 [0.750 to 6.03] | 2.00 [0.500 to 4.00] | 1.50 [0.500 to 3.50] | 2.50 [1.00 to 8.03] | 2.00 [0.500 to 8.00]

5. Secondary Outcome: Plasma Decay Half-Life (t1/2) of Prazosin
Description: Plasma terminal elimination half-life of Prazosin was measured.
Time Frame: 0 (pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 10, 12, 24 hours post-dose on Day 1 of each period
Population: The t1/2 analysis population is defined as all participants randomized and treated who had at least 1 of the PK parameters of secondary interest in at least 1 treatment period.
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Prazosin HCL 1x2 mg (Barceloneta) | Prazosin HCL 1x2 mg (Ascoli) | Prazosin HCL 2x1 mg (Ascoli) | Prazosin HCL 1x5 mg (Barceloneta) | Prazosin HCL 1x5 mg (Ascoli)
Number analyzed (Participants) | 31 | 32 | 31 | 32 | 33
hr | 5.330 (1.2494) | 5.236 (1.0565) | 5.022 (1.1691) | 4.676 (1.1422) | 4.775 (1.1594)

6. Secondary Outcome: Number of Participants With Adverse Events (AEs) According to Seriousness
Description: Adverse events (AEs): any untoward medical occurrence in a clinical investigation participant administered a product or medical device, without regard to causality. Treatment-emergent AEs (TEAEs): AEs which occurred for the first time during the effective duration of treatment or AEs that increased in severity during treatment. Serious AEs (SAEs) were any untoward medical occurrence at any dose that resulted in death; was life-threatening; required inpatient hospitalization or caused prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity (substantial disruption of the ability to conduction normal life functions). Time frame for safety monitoring was from screening to Follow-Up Completion (Day 35 after the last dose administration of the last period), and the actual time frame might vary according to the number of doses received and the length of washing period of each dose for each participant.
Time Frame: Time frame varied from 20 days to 94 days for cohort 1, and 8 days to 73 days for cohort 2.
Population: All participants randomly assigned to study intervention and who had at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Prazosin HCL 1x2 mg (Barceloneta) | Prazosin HCL 1x2 mg (Ascoli) | Prazosin HCL 2x1 mg (Ascoli) | Prazosin HCL 1x5 mg (Barceloneta) | Prazosin HCL 1x5 mg (Ascoli)
Number analyzed (Participants) | 34 | 33 | 33 | 33 | 34
Participants
  Participants with non-serious AEs (all-causality) | 10 | 5 | 6 | 17 | 18
  Participants with non-serious AEs (treatment-related) | 9 | 4 | 5 | 16 | 18
  Participants with SAEs (all-causality) | 1 | 0 | 0 | 0 | 0
  Participants with SAEs (treatment-related) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Time frame for safety monitoring was from screening to Follow-Up Completion (Day 35 after the last dose administration of the last period), and the actual time frame might vary according to the number of doses received and the length of washing period of each dose for each participant. Actual time frame varied from 20 days to 94 days for cohort 1, and 8 days to 73 days for cohort 2.
Description: All participants were included in adverse event monitoring whether they received study treatment or not, and for the AE reporting, AEs (all-cause mortality, serious adverse events, other adverse events) were reported by study treatments that the participants received.
Arm/Group | Prazosin HCL 1x2 mg (Barceloneta) | Prazosin HCL 1x2 mg (Ascoli) | Prazosin HCL 2x1 mg (Ascoli) | Prazosin HCL 1x5 mg (Barceloneta) | Prazosin HCL 1x5 mg (Ascoli)
All-Cause Mortality (participants affected / at risk) | 1/34 | 0/33 | 0/33 | 0/33 | 0/34
Serious Adverse Events (participants affected / at risk) | 1/34 | 0/33 | 0/33 | 0/33 | 0/34
Other Adverse Events (participants affected / at risk) | 8/34 | 4/33 | 5/33 | 16/33 | 18/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prazosin HCL 1x2 mg (Barceloneta) (N=34) | Prazosin HCL 1x2 mg (Ascoli) (N=33) | Prazosin HCL 2x1 mg (Ascoli) (N=33) | Prazosin HCL 1x5 mg (Barceloneta) (N=33) | Prazosin HCL 1x5 mg (Ascoli) (N=34)
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Prazosin HCL 1x2 mg (Barceloneta) (N=34) | Prazosin HCL 1x2 mg (Ascoli) (N=33) | Prazosin HCL 2x1 mg (Ascoli) (N=33) | Prazosin HCL 1x5 mg (Barceloneta) (N=33) | Prazosin HCL 1x5 mg (Ascoli) (N=34)
Nausea (Gastrointestinal disorders) | 2 | 1 | 1 | 7 | 9
Headache (Nervous system disorders) | 2 | 2 | 2 | 3 | 5
Orthostatic hypotension (Vascular disorders) | 4 | 1 | 2 | 3 | 2
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 4
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 9 | 7
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-02-22): https://cdn.clinicaltrials.gov/large-docs/43/NCT04967443/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-05): https://cdn.clinicaltrials.gov/large-docs/43/NCT04967443/SAP_001.pdf